CLINICAL TRIAL: NCT04429360
Title: What is the Effect of Prolapse Surgery on Voiding?
Acronym: PROVOID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Prof Yves Jacquemyn, Head of Department Gynecology, UZA, Universiteit Antwerpen
Other Study IDs: EDGE000835
Record Dates: First submitted 2020-04-30; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Pelvic Organ Prolapse; Stress Urinary Incontinence; Overactive Bladder; Voiding Disorders; Urge Incontinence
Keywords: Pelvic Organ Prolapse; Surgery; 3D/4D imaging; urinary incontinence; voiding dysfunction; patient reported outcome
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress; Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pelvic reconstructive surgery — Pelvic reconstructive surgery

SUMMARY:
The aim of our study is to examine the effect of prolapse surgery on voiding. Our study is the very first one to combine several innovative low-invasive and low-cost methods to analyse the amelioration or deterioration of voiding function after surgery for pelvic organ prolapse using 3D/4D translabial ultrasound, home-uroflowmetry and patient reported quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* Dutch, French or English- speaking women
* symptoms of pelvic organ prolapse
* preoperatively pelvic floor surgery.

Exclusion Criteria:

- history of neurological disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women attending a gynecological unit with symptoms of pelvic organ prolapse and who will undergo pelvic floor surgery as management of their symptoms.
Sampling Method: Probability Sample
Enrollment: 453 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-06-08 (Estimated); Study Completion 2023-06-08 (Estimated)

PRIMARY OUTCOMES:
Change in lower urinary tract symptoms pre- postoperatively | 1 year follow-up
  Voiding diary
Change in lower urinary tract symptoms pre- postoperatively | 1 year follow-up
  Questionnaire: PFDI-20

SECONDARY OUTCOMES:
Change in clinical outcome measures | 1 year follow-up
  POP-Q
Change in clinical outcome measures | 1 year follow-up
  Transperineal ultrasound (TPUS)
Change in voiding | 1 year follow-up
  home-uroflowmetry
Change in QoL | 1 year follow-up
  Questionnaire: PFIQ-7
Change in QoL | 1 year follow-up
  Questionnaire: PISQ-12

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No